CLINICAL TRIAL: NCT05972057
Title: A Prediction Model of Long-term Postoperative Cognitive Dysfunction and Delirium After Cardiac Surgery Based on Peripheral Blood Biomarkers： A Prospective Cohort Study(PPSB)
Brief Title: Prediction Model of Long-term Cognitive Dysfunction and Delirium After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PPSB
Record Dates: First submitted 2023-04-06; First posted 2023-08-02 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Delirium; Cognitive Dysfunction
MeSH Terms: conditions — Delirium; Cognitive Dysfunction | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac surgery — All cardiac surgery patients who met the inclusion criteria were included in the cardiac surgery department of Renji Hospital.

SUMMARY:
Delirium is a clinical syndrome caused by normal dysfunction of the brain, characterized by reduced awareness and responsiveness to the environment, as well as orientation disorders, incoherent thinking and memory disorders. Delirium indicates poor recovery of cognitive function, decreased ability of daily life, may need to enter nursing homes, and even lead to adverse outcomes such as death. According to a number of clinical studies, middle-aged and elderly people are prone to delirium after undergoing major surgery. Delirium occurs in 31 % -40 % of patients over 50 years old after cardiac surgery. Compared with patients without postoperative delirium, patients with postoperative delirium had significant cognitive impairment within 1 year after cardiac surgery. The occurrence of delirium suggests that the patient 's brain has become fragile, cognitive function has begun to decline, and the risk of future dementia has increased.

Secondly, delirium and dementia have overlapping clinical features and common pathogenic mechanisms. Some scholars even speculate that delirium and dementia represent different stages of a common process. It is generally believed that the peripheral immune system may be involved in the pathogenesis and progression of dementia through the dysfunctional blood-brain barrier. The activation of microglia and astrocytes leads to the release of chemokines, which can recruit peripheral immune cells to the central nervous system. At the same time, cytokines released by peripheral cells can cross the blood-brain barrier and act on glial cells to change their phenotype.

This study is a prospective cohort study of patients aged 65 and over who are about to undergo elective cardiac surgery.CyTOF can achieve accurate immunophenotyping of cell populations while comprehensively and accurately detecting and analyzing cytokines and signaling pathways. Therefore, the detection of peripheral blood biomarkers may effectively predict the risk of long-term cognitive dysfunction and postoperative delirium in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Patients undergoing elective cardiac surgery with cardiopulmonary bypass
* Sign informed consent

Exclusion Criteria:

* serious dementia, encephalopathy, mental illness or other neurological diseases
* Patients who could not take neurocognitive tests due to other reasons ( such as language, hearing or visual impairment )
* Patients with stage 3 or 4 malignant tumors, and patients with pancreatic cancer, gallbladder cancer, cholangiocarcinoma and other tumors with high malignancy and expected survival time less than 1 year
* American Society of Anesthesiologists ( ASA ) classification IV or V patients

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: During the implementation of the project, all patients with cardiac surgery who met the inclusion criteria were included in the Department of Cardiac Surgery of Renji Hospital. The total sample size was the sum of all patients by the project deadline.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-29 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium | up to 5 days after surgery
  To establish a risk factor prediction model for postoperative delirium in patients aged 65 and over undergoing elective cardiac surgery by detecting peripheral blood biomarkers by CyTOF.

SECONDARY OUTCOMES:
long-term cognitive dysfunction | 1 year after surgery
  To establish a risk factor prediction model for long-term cognitive impairment in patients aged 65 and over undergoing elective cardiac surgery by detecting peripheral blood biomarkers by CyTOF.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China